CLINICAL TRIAL: NCT00315497
Title: Longitudinal Protocol for Giant Cell Arteritis
Brief Title: Determining Disease Activity Biomarkers in Individuals With Giant Cell Arteritis
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Office of Rare Diseases (ORD) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Rare Diseases Clinical Research Network (Network)
Responsible Party: Principal Investigator, Peter Merkel, Professor, University of Pennsylvania
Other Study IDs: VCRC5502; U54AR057319 (NIH)
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Temporal Arteritis
Keywords: Giant Cell Arteritis
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (serum and plasma), urine, and DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Giant cell arteritis (GCA), also known as temporal arteritis, is a disease that usually only occurs in older adults. GCA causes inflammation of blood vessels, or vasculitis. In order to properly treat this disease, it is critical that the level of disease activity can be determined over the course of the disease. The purpose of this study is to determine new biological markers, or biomarkers, that may be used to assess the severity of disease in people with GCA.

DETAILED DESCRIPTION:
GCA is a rare autoimmune disorder and is the most common type of inflammation of medium- to large-sized blood vessels in the body. It usually only occurs in older adults. The most common symptoms of GCA include headache, pain in the shoulders and hips (polymyalgia rheumatica), pain in the jaw (jaw claudication), fever, and blurred vision. Organ-specific markers of injury or damage as well as direct markers of vascular damage and inflammation are currently used by clinicians to assess GCA disease progression; however, these markers are not very useful in guiding treatment. There are also blood tests that clinicians use to monitor GCA activity, such as erythrocyte sedimentation rate (ESR) and C-reactive protein (CRP), but these tests lack specificity and sensitivity. Most treatments available now for GCA are toxic, therefore if other markers indicating disease activity can be found, it may lead to the development of less toxic treatments. This study will use new scientific methods to identify new biomarkers that can be used to monitor disease activity in GCA patients. These biomarkers may be used to help direct clinical care for GCA patients and assist in future drug development.

Study visits will occur monthly for the first year, then every 3 months thereafter for the remainder of the study. Blood and urine collection will occur at every visit. A physical exam and medical and medication history will occur every 3 months; also, participants will be asked to complete several questionnaires to assess disease activity, health status, and tobacco, alcohol, and drug use. Participants may have additional study visits if a disease flare or disease-related complications occur during the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GCA, meeting at least 3 of the following 5 American College of Rheumatology (ACR) criteria for the diagnosis of GCA:

  1. At least 50 years of age at disease onset
  2. New onset or new type of localized pain in the head
  3. Temporal artery abnormality (i.e., temporal artery tenderness to palpation or decreased pulsation unrelated to arteriosclerosis of cervical arteries)
  4. ESR of greater than 40 mm in the first hour by the Westergren method
  5. Temporal artery biopsy showing vasculitis characterized by a predominance of mononuclear cell infiltration or granulomatous inflammation, usually with multinucleated giant cells

Exclusion Criteria:

* Unable to give informed consent and sign the consent form

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with giant cell arteritis. Enrollment will be sequential and participants will have disease in various stages and of different duration.
Sampling Method: Non-Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Discover biomarkers in Giant cell arteritis capable of measuring disease activity and response to treatment. | Study completion

SECONDARY OUTCOMES:
Measure the predictive value of biomarkers for clinical outcome in Giant cell arteritis. | Study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. Merkel, MD, MPH, Study Chair — University of Pennsylvania
Locations (9):
- United States (7):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - Mayo Clinic College of Medicine, Rochester, Minnesota
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Canada (2):
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonzalez-Gay MA, Amoli MM, Garcia-Porrua C, Ollier WE. Genetic markers of disease susceptibility and severity in giant cell arteritis and polymyalgia rheumatica. Semin Arthritis Rheum. 2003 Aug;33(1):38-48. doi: 10.1053/sarh.2002.50025. PMID 12920695
- [Background] Goronzy JJ, Weyand CM. Cytokines in giant-cell arteritis. Cleve Clin J Med. 2002;69 Suppl 2:SII91-4. doi: 10.3949/ccjm.69.suppl_2.sii91. PMID 12086274
- [Background] Weyand CM, Fulbright JW, Hunder GG, Evans JM, Goronzy JJ. Treatment of giant cell arteritis: interleukin-6 as a biologic marker of disease activity. Arthritis Rheum. 2000 May;43(5):1041-8. doi: 10.1002/1529-0131(200005)43:53.0.CO;2-7. PMID 10817557
- [Background] Weyand CM, Goronzy JJ. Giant-cell arteritis and polymyalgia rheumatica. Ann Intern Med. 2003 Sep 16;139(6):505-15. doi: 10.7326/0003-4819-139-6-200309160-00015. PMID 13679329
- See also: Vasculitis Clinical Research Network — https://www.rarediseasesnetwork.org/cms/vcrc/
- See also: Rare Disease Clinical Research Network — https://www.rarediseasesnetwork.org/